CLINICAL TRIAL: NCT00723255
Title: A Phase II Evaluation of Combination Bevacizumab (NCI-Supplied Agent: NSC #70486) and Temsirolimus (CCI-779, NCI-Supplied Agent, NSC #683864) in the Treatment of Recurrent or Persistent Endometrial Carcinoma
Brief Title: Bevacizumab and Temsirolimus in Treating Patients With Recurrent or Persistent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00598; NCI-2009-00598 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000601291; GOG-0229G (Other: Gynecologic Oncology Group); GOG-0229G (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2008-07-25; First posted 2008-07-28 (Estimated); Results first posted 2015-08-05 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Recurrent Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Bevacizumab; temsirolimus; Sirolimus

ARMS (1):
- Treatment (bevacizumab, temsirolimus) (Experimental): Patients receive bevacizumab IV on days 1 and 15 and temsirolimus IV on days 1, 8, 15, and 22.
  Interventions: Biological: bevacizumab; Drug: temsirolimus

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel

SUMMARY:
This phase II trial is studying the side effects of giving bevacizumab together with temsirolimus and to see how well it works in treating patients with recurrent or persistent endometrial cancer. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for their growth. Giving bevacizumab together with temsirolimus may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the activity of bevacizumab and temsirolimus, in terms of 6-month progression-free survival (PFS) and objective tumor response, in patients with recurrent or persistent endometrial cancer.

II. To determine the nature and degree of toxicity of this regimen in these patients.

SECONDARY OBJECTIVES:

I. To determine the duration of PFS and overall survival of patients treated with this regimen.

II. To determine the effects of prognostic factors (i.e., performance status, histological subtype, and grade) in patients treated with this regimen.

TERTIARY OBJECTIVES:

I. To compare the proportion of patients with objective tumor response and PFS at 6 months receiving the combination of bevacizumab and temsirolimus with those for the single agents bevacizumab and temsirolimus using historical controls.

OUTLINE: This is a multicenter study.

Patients receive bevacizumab IV on days 1 and 15 and temsirolimus IV on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 3 months for 2 years, then every 6 months for 3 years, for a total of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed endometrial carcinoma (from primary tumor) including any of the following cell types:

  * Endometrioid adenocarcinoma
  * Serous adenocarcinoma
  * Undifferentiated carcinoma
  * Clear cell adenocarcinoma
  * Mixed epithelial carcinoma
  * Adenocarcinoma not otherwise specified
  * Mucinous adenocarcinoma
  * Squamous cell carcinoma
  * Transitional cell carcinoma
  * Mesonephric carcinoma
* Recurrent or persistent disease that is refractory to curative therapy or established treatments
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* Must have ≥ 1 target lesion to assess response as defined by RECIST

  * Tumors within a previously irradiated field are designated as "non-target" lesions in the absence of documented disease progression or a biopsy to confirm persistence for ≥ 90 days after completion of radiotherapy
* Must have received 1 prior chemotherapeutic regimen for management of endometrial carcinoma

  * May have received 1 additional cytotoxic regimen for management of this disease
* Not eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, including any active GOG Phase III protocol for patients with endometrial carcinoma
* No history or evidence of CNS disease, including primary brain tumor or any brain metastases upon physical examination
* GOG performance status (PS) 0-2 (for patients who have received 1 prior regimen) OR PS 0-1 (for patients who have received 2 prior regimens)
* ANC ≥ 1,500/mcL
* Platelet count ≥ 100,000/mcL
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Urine protein:creatinine ratio < 1.0 OR urine protein < 1,000 mg by 24-hour urine collection
* INR ≤ 1.5 OR in-range INR between 2 and 3 if patient is on a stable dose of therapeutic warfarin
* PTT ≤ 1.5 times ULN
* Fasting cholesterol < 350 mg/dL
* Fasting triglycerides < 400 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Seizures allowed provided they are controlled with standard medical therapy
* No active infection requiring antibiotics, except uncomplicated urinary tract infection
* No active bleeding or pathologic conditions that carry high risk of bleeding, (e.g., known bleeding disorder, coagulopathy, or tumor involving major vessels)
* No serious, non-healing wound, ulcer, or bone fracture, including abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 3 months

  * No prior underlying lesions that caused the fistula or perforation that have not been corrected
* No prior interstitial pneumonitis
* No clinically significant cardiovascular disease, including any of the following:

  * Uncontrolled hypertension, defined as systolic blood pressure (BP) > 150 mm Hg or diastolic BP > 90 mm Hg
  * Myocardial infarction or unstable angina within the past 6 months
  * New York Heart Association class II-IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Peripheral vascular disease ≥ grade 2
* No cerebrovascular accident, transient ischemic attack, or subarachnoid hemorrhage within the past 6 months
* No uncontrolled diabetes

  * Hemoglobin A1C < 10
* No other invasive malignancies within the past 5 years, except nonmelanoma skin cancer and other specific malignancies (e.g., localized breast, head and neck, or skin cancer that completed treatment > 3 years prior to study and remain disease-free)
* No significant traumatic injury within the past 28 days
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies
* Concurrent prophylactic or therapeutic anticoagulation* (e.g., warfarin) allowed
* Recovered from recent surgery, radiotherapy, or chemotherapy
* No prior bevacizumab or other VEGF pathway-targeted therapy
* No prior temsirolimus, everolimus, deforolimus, sirolimus, or any other mTor/PI3K pathway-targeted therapy
* No prior non-cytotoxic chemotherapy for management of this disease, except hormonal therapy

  * At least 1 week since prior hormonal therapy directed at the malignant tumor
* No prior therapy that contraindicates this protocol therapy
* No prior radiotherapy to any portion of the abdominal cavity or pelvis within the past 5 years, except treatment of endometrial cancer

  * Prior radiotherapy for localized cancer of the breast, head and neck, or skin is allowed, provided it was completed > 3 years prior to study entry and patient remains free of recurrent or metastatic disease
* No prior chemotherapy for any abdominal or pelvic tumor within the past 5 years, except treatment of endometrial cancer

  * Prior adjuvant chemotherapy for localized breast cancer allowed, provided it was completed > 3 years prior to study entry and the patient remains free of recurrent or metastatic disease
* Prior treatment with an anthracycline (i.e., doxorubicin and/or liposomal doxorubicin) allowed provided ejection fraction < 50%
* More than 28 days since prior major surgery or open biopsy
* More than 7 days since minor surgical procedures, fine needle aspirates, or core biopsies
* At least 3 weeks since prior therapy directed at the malignant tumor, including immunologic agents
* No concurrent major surgery
* No concurrent prophylactic filgrastim (G-CSF) or thrombopoietic agents
* No concurrent amifostine or other protective reagents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-09; Primary Completion 2011-07-15 (Actual); Study Completion 2016-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Alvarez, Principal Investigator — Gynecologic Oncology Group
Locations (41):
- United States (41):
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Memorial University Medical Center, Savannah, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University Medical Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Services, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Gynecologic Oncology of West Michigan PLLC, Grand Rapids, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Ozark Health Ventures LLC-Cancer Research for The Ozarks Springfield, Springfield, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Women's Cancer Care Associates LLC, Albany, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Gynecologic Oncology Network, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 9/8/2008 and closed to accrual on 3/22/2010 (and was suspended from 1/19/2009 to 12/7/2009).
Groups:
- Bevacizumab Plus Temsirolimus: Bevacizumab 10 mg/kg IV every other week plus Temsirolimus 25 mg IV weekly (one cycle = 4 weeks) until disease progression or adverse effects prohibit further therapy
Period: Overall Study
Arm/Group | Bevacizumab Plus Temsirolimus
Started | 53
Completed | 49 (Eligible and treated patients)
Not Completed | 4
Not completed — Ineligible: Inadequate pathology | 1
Not completed — Ineligible: Second primary | 1
Not completed — Ineligible: Wrong Primary | 2

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab Plus Temsirolimus
Number analyzed (Participants) | 49
Age, Customized [Number; unit: participants]
  20-29 years | 0
  30-39 years | 1
  40-49 years | 4
  50-59 years | 11
  60-69 years | 21
  70-79 years | 11
  80-89 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Complete and Partial Tumor Response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.0
Time Frame: Scans are done while patient is on study therapy every other cycle for the first 6 months; then every 3 cycles thereafter; and at any other time if clinically indicated based on symptoms or physical signs suggestive of progressive disease
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab Plus Temsirolimus
Number analyzed (Participants) | 49
percentage of participants | 24.5 [14.8 to 36.6]

2. Primary Outcome: Progression-free Survival at 6 Months
Description: Percentage of patients who are progression-free 6 months after study entry. Progression-Free Survival is the period from study entry until disease progression, death or date of last contact.
Time Frame: Every other cycle for 6 months
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab Plus Temsirolimus
Number analyzed (Participants) | 49
percentage of participants | 46.9 [34.6 to 59.6]

3. Primary Outcome: Frequency and Severity of Adverse Events Assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Time Frame: Every cycle and 30 days after the last treatment, an average of 5 years.
Population: Eligible and evaluable patients
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1 (CTCAE v 3.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria version 3.0
- Grade 2 (CTCAE v 3.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria version 3.0
- Grade 3 (CTCAE v 3.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria version 3.0
- Grade 4 (CTCAE v 3.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria version 3.0
- Grade 5 (CTCAE v 3.0): Number of patients who experienced a grade 5 event using Common Terminology Criteria version 3.0
Arm/Group | Grade 0 | Grade 1 (CTCAE v 3.0) | Grade 2 (CTCAE v 3.0) | Grade 3 (CTCAE v 3.0) | Grade 4 (CTCAE v 3.0) | Grade 5 (CTCAE v 3.0)
Number analyzed (Participants) | 49 | 49 | 49 | 49 | 49 | 49
Participants
  Leukopenia | 20 | 13 | 15 | 1 | 0 | 0
  Thrombocytopenia | 24 | 18 | 4 | 3 | 0 | 0
  Neutropenia | 28 | 7 | 9 | 5 | 0 | 0
  Anemia | 14 | 17 | 14 | 3 | 1 | 0
  Other hematologic | 46 | 1 | 2 | 0 | 0 | 0
  Allergy/immunology | 47 | 1 | 1 | 0 | 0 | 0
  Cardiac | 33 | 3 | 7 | 5 | 1 | 0
  Coagulation | 48 | 0 | 0 | 1 | 0 | 0
  Constitutional | 12 | 9 | 18 | 9 | 1 | 0
  Dermatologic | 18 | 13 | 16 | 2 | 0 | 0
  Endocrine | 48 | 1 | 0 | 0 | 0 | 0
  Gastrointestinal | 5 | 11 | 15 | 17 | 1 | 0
  Genitourinary/renal | 44 | 3 | 1 | 1 | 0 | 0
  Hemorrhage | 25 | 22 | 1 | 1 | 0 | 0
  Infection | 34 | 0 | 8 | 6 | 0 | 1
  Lymphatics | 40 | 5 | 3 | 1 | 0 | 0
  Metabolic | 9 | 11 | 12 | 14 | 3 | 0
  Musculoskeletal | 43 | 3 | 2 | 1 | 0 | 0
  Neurosensory | 43 | 5 | 1 | 0 | 0 | 0
  Other neurological | 41 | 4 | 3 | 1 | 0 | 0
  Ocular/visual | 45 | 2 | 1 | 1 | 0 | 0
  Pain | 18 | 12 | 10 | 8 | 1 | 0
  Pulmonary | 26 | 14 | 7 | 1 | 0 | 1
  Sexual/reproductive | 48 | 1 | 0 | 0 | 0 | 0
  Vascular | 47 | 0 | 0 | 1 | 1 | 0
  Death, not CTC coded | 48 | 0 | 0 | 0 | 0 | 1

4. Secondary Outcome: Progression-Free Survival
Description: Progression-Free Survival is the period from study entry until disease progression, death or date of last contact.
Time Frame: as for outcome 1
Population: Eligible and Treated Patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab Plus Temsirolimus
Number analyzed (Participants) | 49
Months | 5.6 [4.0 to 7.7]

5. Secondary Outcome: Overall Survival
Description: The observed length of life from entry into the study to death or the date of last contact.
Time Frame: From entry into the study to death or the date of last contact, up to 5 years
Population: Eligible and Treated Patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab Plus Temsirolimus
Number analyzed (Participants) | 49
Months | 16.9 [10.7 to 21.2]

6. Secondary Outcome: Complete and Partial Tumor Response by RECIST 1.0 by Performance Status
Description: Complete and Partial Tumor Response by RECIST 1.0
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Performance Status 0: Patients with performance status 0 Performance Status 0: Fully active, able to carry on all pre-disease performance without restriction
- Performance Status 1,2: Patients with performance status 1 or 2 Performance Status 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light house work Performance Status 2: Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours
Arm/Group | Performance Status 0 | Performance Status 1,2
Number analyzed (Participants) | 29 | 20
percentage of participants | 24 [10 to 44] | 25 [9 to 49]

7. Secondary Outcome: Progression-free Survival at 6 Months by Performance Status
Description: as for outcome 2
Time Frame: Every other cycle for 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Performance Status 0 | Performance Status 1,2
Number analyzed (Participants) | 29 | 20
percentage of participants | 48 [29 to 67] | 45 [23 to 68]

8. Secondary Outcome: Complete and Partial Tumor Response by RECIST 1.0 by Histologic Type
Description: Complete and Partial Tumor Response by RECIST 1.0
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Endometrioid Adenocarcinoma: Patients with endometrioid adenocarcinoma
- Other Histologic Types: Patients with other histologic types, including benign (not otherwise specified) (n=1), unspecified adenocarcinoma (n=1), clear cell carcinoma (n=2), mucinous adenocarcinoma (n=1), mixed epithelial carcinoma (n=5), undifferentiated carcinoma (n=1), serous adenocarcinoma (n=4)
Arm/Group | Endometrioid Adenocarcinoma | Other Histologic Types
Number analyzed (Participants) | 34 | 15
percentage of participants | 21 [9 to 38] | 33 [12 to 62]

9. Secondary Outcome: Progression-free Survival at 6 Months by Histologic Type
Description: as for outcome 2
Time Frame: Every other cycle for 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Endometrioid Adenocarcinoma | Other Histologic Types
Number analyzed (Participants) | 34 | 15
percentage of participants | 44 [27 to 62] | 53 [27 to 79]

10. Secondary Outcome: Complete and Partial Tumor Response by RECIST 1.0 by Tumor Grade
Description: Complete and Partial Tumor Response by RECIST 1.0
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Grade 1,2: Patients with grade 1-2 tumors (patients with missing grade excluded, n=7)
- Grade 3: Patients with grade 3 tumors (patients with missing grade excluded, n=7)
Arm/Group | Grade 1,2 | Grade 3
Number analyzed (Participants) | 20 | 15
percentage of participants | 30 [12 to 54] | 18 [5 to 40]

11. Secondary Outcome: Progression-free Survival at 6 Months by Tumor Grade
Description: as for outcome 2
Time Frame: Every other cycle for 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Grade 1,2 | Grade 3
Number analyzed (Participants) | 20 | 15
percentage of participants | 60 [36 to 81] | 32 [14 to 55]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) during treatment (up to 30 days after treatment completion). All Serious Adverse Events (SAEs) up to 30 days after treatment completion and considered to be treatment related between 30 days and 5 years after treatment completion.
Arm/Group | Bevacizumab Plus Temsirolimus
Serious Adverse Events (participants affected / at risk) | 31/49
Other Adverse Events (participants affected / at risk) | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab Plus Temsirolimus (N=49)
Hypertension (Cardiac disorders) | 1
Lt Ventricular Systolic Dysfunction (Cardiac disorders) | 1
Inr (Vascular disorders) | 1
Fever (General disorders) | 1
Death No Ctcae Term - Sudden Death (General disorders) | 2
Fistula, Gi - Rectum (Gastrointestinal disorders) | 1
Obstruction, Gi - Colon (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 2
Perforation, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Anorexia (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 1
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Dental-Tooth (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 1
Proteinuria (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 1
Pain: Neck (General disorders) | 1
Pain: Rectum (General disorders) | 2
Pain: Abdominal Pain Nos (General disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Obstruction, Gu - Ureter (Renal and urinary disorders) | 1
Fistula, Gu - Vagina (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab Plus Temsirolimus (N=49)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 2
Rhinitis (Immune system disorders) | 3
Tinnitus (Ear and labyrinth disorders) | 4
Neutrophils (Blood and lymphatic system disorders) | 23
Platelets (Blood and lymphatic system disorders) | 27
Leukocytes (Blood and lymphatic system disorders) | 29
Lymphopenia (Blood and lymphatic system disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 39
Palpitations (Cardiac disorders) | 2
S/N Arrhythmia: Sinus Tachycardia (Cardiac disorders) | 4
Vasovagal Episode (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 15
Restrictive Cardiomyopathy (Cardiac disorders) | 1
Cardiac General - Other (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 2
Inr (Vascular disorders) | 1
Ptt (Vascular disorders) | 1
Constitutional Symptoms - Other (General disorders) | 1
Fever (General disorders) | 7
Weight Loss (General disorders) | 16
Rigors/Chills (General disorders) | 2
Fatigue (General disorders) | 38
Insomnia (General disorders) | 5
Death No Ctcae Term - Disease Progression Nos (General disorders) | 2
Nail Changes (Skin and subcutaneous tissue disorders) | 10
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 12
Bruising (Skin and subcutaneous tissue disorders) | 4
Acne (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 24
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Decubitus (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 10
Burn (Skin and subcutaneous tissue disorders) | 1
Flushing (Skin and subcutaneous tissue disorders) | 3
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Ulceration (Skin and subcutaneous tissue disorders) | 3
Hot Flashes (Endocrine disorders) | 4
Hypothyroidism (Endocrine disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Fistula, Gi - Rectum (Gastrointestinal disorders) | 1
Ulcer,gi - Stoma (Gastrointestinal disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 4
Heartburn (Gastrointestinal disorders) | 2
Mucositis (Functional/Sympt) - Pharynx (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 6
Distention (Gastrointestinal disorders) | 1
Taste Alteration (Gastrointestinal disorders) | 10
Incontinence, Anal (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 1
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 16
Mucositis (Clinical Exam) - Stomach (Gastrointestinal disorders) | 1
Perforation, Gi - Small Bowel Nos (Gastrointestinal disorders) | 2
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 17
Mucositis (Clinical Exam) - Anus (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 20
Anorexia (Gastrointestinal disorders) | 21
Dehydration (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 20
Nausea (Gastrointestinal disorders) | 29
Diarrhea (Gastrointestinal disorders) | 29
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 3
Hemorrhage, Gu - Vagina (Vascular disorders) | 3
Hemorrhage, Gi - Rectum (Vascular disorders) | 7
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 23
Hematoma (Vascular disorders) | 1
Hemorrhage, Gi - Anus (Vascular disorders) | 1
Hemorrhage, Gi - Colon (Vascular disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Nose (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 3
Inf W/Nml Or Gr 1 Or 2 Anc: Dental-Tooth (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 7
Inf W/Nml Or Gr 1 Or 2 Anc: Abdomen Nos (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Ungual (Nails) (Infections and infestations) | 1
Infection - Other (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bronchus (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Sinus (Infections and infestations) | 2
Inf Unknown Anc: External Ear (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 3
Edema: Limb (Blood and lymphatic system disorders) | 11
Edema: Head And Neck (Blood and lymphatic system disorders) | 2
Ast (Metabolism and nutrition disorders) | 14
Gfr (Metabolism and nutrition disorders) | 2
Cholesterol,serum High (Metabolism and nutrition disorders) | 28
Proteinuria (Metabolism and nutrition disorders) | 1
Creatinine (Metabolism and nutrition disorders) | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 10
Alt (Metabolism and nutrition disorders) | 13
Alkaline Phosphatase (Metabolism and nutrition disorders) | 5
Bilirubin (Metabolism and nutrition disorders) | 2
Lipase (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 12
Hyponatremia (Metabolism and nutrition disorders) | 12
Hypertriglyceridemia (Metabolism and nutrition disorders) | 27
Cpk (Metabolism and nutrition disorders) | 1
Bicarbonate, Serum-Low (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 14
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 20
Hypokalemia (Metabolism and nutrition disorders) | 17
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 12
Fibrosis-Deep Connective Tissue (Musculoskeletal and connective tissue disorders) | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 9
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 5
Mood Alteration - Depression (Nervous system disorders) | 7
Mood Alteration - Anxiety (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Cognitive Disturbance (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 2
Memory Impairment (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 6
Neuropathy-Sensory (Nervous system disorders) | 18
Neuropathy-Motor (Nervous system disorders) | 2
Watery Eye (Eye disorders) | 2
Cataract (Eye disorders) | 1
Flashing Lights/Floaters (Eye disorders) | 3
Blurred Vision (Eye disorders) | 8
Pain: Urethra (General disorders) | 1
Pain: Perineum (General disorders) | 1
Pain: Pelvis (General disorders) | 1
Pain: Vagina (General disorders) | 1
Pain: Chest Wall (General disorders) | 1
Pain: Throat/Pharynx/Larynx (General disorders) | 3
Pain: Larynx (General disorders) | 1
Pain: Head/Headache (General disorders) | 15
Pain: Extremity-Limb (General disorders) | 7
Pain: Back (General disorders) | 4
Pain: Joint (General disorders) | 12
Pain: Bone (General disorders) | 3
Pain: Bladder (General disorders) | 3
Pain: Pain Nos (General disorders) | 1
Pain: Stomach (General disorders) | 1
Pain: Rectum (General disorders) | 3
Pain: Oral Cavity (General disorders) | 2
Pain: Dental/Teeth/Peridontal (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 17
Pain: Scalp (General disorders) | 1
Pain: Oral - Gums (General disorders) | 1
Pain: Middle Ear (General disorders) | 3
Pain: External Ear (General disorders) | 1
Pain: Face (General disorders) | 1
Pain: Muscle (General disorders) | 3
Pain: Anus (General disorders) | 1
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 1
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 3
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 18
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18
Cystitis (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Obstruction, Gu - Ureter (Renal and urinary disorders) | 1
Incontinence, Urinary (Renal and urinary disorders) | 1
Fistula, Gu - Vagina (Renal and urinary disorders) | 1
Bladder Spasm (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 9
Vaginitis (Reproductive system and breast disorders) | 1
Vaginal Discharge (Reproductive system and breast disorders) | 1
Flu-Like Syndrome (General disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less